CLINICAL TRIAL: NCT02721342
Title: Remission Clinic: Computed Registry for the Ambulatory Follow up of Patients With Proteinuric Chronic Nephropathies Treated Based on a Standard Multipharmacological Model Aimed at Normalizing Proteinuria and Stabilizing the Renal Function
Brief Title: Remission Clinic in Proteinuric Chronic Nephropathies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: Remission Clinic
Record Dates: First submitted 2016-03-14; First posted 2016-03-29 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic proteinuric nephropathies
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Ramipril; Irbesartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ramipril, Irbesartan and Atorvastin treatment: A multidrug approach, including Angiotensin II Converting Enzyme (ACE) inhibitor, Ramipril, and Angiotensin II Receptor Blocker (ARB), Irbesartan, and Atorvastin will be done. Treatment doses of drugs will be up-titrated gradually considering the tolerability.
  Interventions: Drug: Ramipril, Irbesartan and Atorvastin

INTERVENTIONS:
Drug: Ramipril, Irbesartan and Atorvastin

SUMMARY:
Most chronic kidney diseases have a progressive evolution characterized by the gradual loss of glomerular filtration rate (GFR), electrolytic imbalance, reduced erythropoietin synthesis and activation of vitamin D. On many occasions, the progressive deterioration of renal function occurs, even when the etiologic factors responsible for the kidney disease are treated and/or eliminated as a result of an auto-sustained mechanism of inflammation and fibrosis. Moreover, chronic nephropathies are often associated with high blood pressure and increased urine protein excretion, being both risk factors of progression toward kidney failure. Many clinical studies have shown the efficacy of antihypertensive therapies, particularly the blockade of renin-angiotensin system, to lower the abnormal urinary protein excretion. Moreover, control of blood pressure and proteinuria slow the rate of renal function decline and in some cases even lead to recovery of kidney function avoiding the need for renal replacement therapies. The set of measures to achieve these results encompasses the term of "renoprotective therapy". However these achievements have been obtained in the setting of clinical trials, and need confirmation in the daily clinical practice.

To this purpose a standardized multidrug intervention model that aims at normalizing the excretion of urinary proteins and stabilizing the renal function has been developed for the outpatient-clinic and named "Remission Clinic".

The applicability of this protocol is aimed for all nephrology and diabetology centers. Through the use of a dedicated database computer network, it will be possible to share clinical, laboratory and treatment data, recorded for each patient enrolled in the Remission Clinic program. With this system, it will be possible to verify if the multidrug approach of the Remission Clinic will allow to improve the clinical course of chronic proteinuric nephropathy. All participants (centers) may access to the Remission Clinic website developed, updated and maintained by the Department of Bioengineering of the Mario Negri Institute, Bergamo, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Proteinuria >0.5 g/24 hours or albuminuria >200 g / min (or >300 g/24 hours) for at least 2 consecutive evaluations regardless of treatment with ACEi and/or ARBs;
* Change in serum creatinine or creatinine clearance less than 30% in the last 3 months;
* No corticosteroids or immunosuppressants at the time of inclusion or given to patient in the last 6 months.

Exclusion Criteria:

* Idiopathic membranous nephropathy;
* Focal segmental glomerulosclerosis;
* Minimal change glomerulopathy;
* Nephritic syndrome;
* Rapidly progressive renal failure (extracapillary glomerulonephritis in active phase);
* Any active renal disease that represents a possible indication to corticosteroids or immunosuppressive therapy;
* Nephropathies secondary to systemic disease susceptible to treatment with corticosteroids or immunosuppressive agents (Systemic Lupus Erythematosus, Vasculitis, Amyloidosis, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic or non-diabetic chronic nephropathies, with no specific contraindications for treatment with ACEi or Sartans.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2009-06; Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Glomerular Filtration Rate (GFR) estimated | Changes from baseline at at least every 3 to 6 months for the duration of the study, an expected average of 10 years.
24 hour proteinuria | Changes from baseline at at least every 3 to 6 months for the duration of the study, an expected average of 10 years.

SECONDARY OUTCOMES:
Number of participants with fatal and non-fatal cardiovascular events | Participants will be followed for the duration of the study, an expected average of 10years.
  Sudden death, myocardial infarction, unstable angina, stroke, transient ischemic attack, lower limb amputation, coronary, carotid or peripheral vessel revascularization.

CONTACTS AND LOCATIONS:
Locations (13):
- Italy (13):
  - Centro di Ricerche Cliniche per le Malattie Rare Aldo e Cele Daccò, Ranica, Bergamo
  - Ospedale Morgagni - Pierantoni - U.O. Nefrologia e Dialisi, Forlì, Forli'
  - Asl 6 Sanluri-P.O. Nostra Signora di Bonaria - U.O. Nefrologia e Dialisi, San Gavino Monreale, Medio Campidano - VS
  - Ospedale C.G. Mazzoni Zona 13 ASUR Marche - U.O. Nefrologia e Dialisi, Ascoli Piceno
  - AORN Moscati - Avellino - U.O. Nefrologia e Dialisi, Avellino
  - A.O. Papa Giovanni XXIII - U.O. Nefrologia e Dialisi, Bergamo
  - A.O. Papa Giovanni XXIII Bergamo - U.O. Diabetologia, Bergamo
  - Azienda Ospedaliera G. Brotzu - U.O. Nefrologia e Dialisi, Cagliari
  - Ospedale Campo di Marte - USL 2 - U.O. Nefrologia, Lucca
  - ARNAS Ospedale Civico Di Cristina Benfratelli - U.O. Nefrologia e Dialisi, Palermo
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Università degli Studi di Palermo - Dipartimento Malattie Cardiovascolari e Nefrourologiche - U.O. Tecniche Dialitiche, Palermo
  - Azienda Ospedaliera Universitaria Pisana - U.O. Nefrologia e Dialisi 2, Pisa
  - Ospedale di Circolo Fondazione Macchi - U.O. Nefrologia e Dialisi, Varese

IPD SHARING:
Plan to Share IPD: No